

## **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH WITH OPTIONAL PROCEDURES

Sleep disturbances in surgical patients with GI cancers: A quantitative and qualitative analysis 2019-1182

| Study Chair: | Sriram Yennu |
|--------------------|-----------------------|
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

#### STUDY SUMMARY

Sleep disturbance (such as difficulty sleeping) is one of the most common complaints of patients after surgery and may affect the ability to carry out daily activities, quality of life, and post-surgery recovery. However, the effects of sleep disturbance have not been studied very much in cancer patients before and after surgery.

The goal of this research study is to collect information about the sleeping habits and health of patients who have gastrointestinal (GI) cancer and who are scheduled for standard of care surgery. Researchers think that if sleep-related symptoms can be diagnosed and managed, the overall symptom burden on patients can be lowered and the overall quality of life can be improved.

## This is an investigational study.

If sleep-related symptoms are identified and managed, your quality of life may improve. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. If you take part in this study, your

NCT05044312 Protocol 2019-1182 May 14, 2020 

appointment times will be longer because of the questionnaires you will complete as part of this study.

You can read a list of potential side effects below in the Possible Risks section of this consent.

Your participation in this study will be over about 30 days after you have been discharged from the hospital.

There is no cost to you for taking part in this study.

You may choose not to take part in this study.

#### 1. STUDY DETAILS

Up to 200 participants will be enrolled in this study. All will take part at MD Anderson.

If you agree to take part in this study, you will have the following tests/procedures performed at the noted time points before surgery, after surgery, and after you are discharged from the hospital. You will sign a separate consent for your standard of care surgery which will explain the procedure and its risks.

Once before the surgery, every day during the 7 days after surgery, at your first post-operative visit (after you are discharged from the hospital), and then at about 30 days after discharge:

- Blood (about 1 teaspoon each time) will be drawn for routine and/or immune system testing. Immune system testing in this study is being done to possibly link sleep disturbances to measurable information (such as immune system testing results).
- You will complete up to 9 questionnaires about your sleep habits, symptoms, and quality of life. It may take up to 30-45 minutes to complete all questionnaires. You will not complete all questionnaires every day.
- You will be given an Actigraph and Fitbit to wear so that researchers can track and measure your activity levels and sleep cycle. You will return the Actigraph to the study team at your first post-operative visit. If you lose, damage, or have technical issues with the Actigraph or Fitbit, tell the study staff right away. The study staff will provide you with a replacement at no cost to you. The study staff may contact you over the phone if there are gaps in data collection through these devices. You will be able to keep the FitBit after you complete the study.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The known side effects are listed in this form, but they will vary

from person to person.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the questionnaire, you are encouraged to contact your doctor or the study chair.

If you are feeling distressed and the study staff or doctor thinks it is needed, you will be referred to another doctor or therapist for additional help.

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Although every effort will be made to keep **study data** safe, there is a chance that your personal health information could be lost or stolen. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

This study may involve unpredictable risks to the participants.

#### OPTIONAL PROCEDURES FOR THE STUDY

You may be asked to take part in the optional procedure below.

**Optional Procedure #1:** If you agree, the study staff will interview you about 5-7 days after your surgery. During the interview, you will be asked about your sleep experience and habits before surgery and if you took any sleep aids, how you slept while you were in the hospital, and how you think your sleeping habits have affected your care and health. The interview should last about 1 hour.

The interview will be audio-recorded and then transcribed (written down). After being transcribed, the audio-recording will be deleted. No patient names will be attached to the interview and if you use names during the interview, they will not be written down.

There are no benefits to you for taking part in the optional procedure. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedure.

## **Optional Procedure Risks**

**Interviews** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the interview, you are encouraged to contact your doctor or the study chair.

## CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES

Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1:** Do you agree to complete the interview after surgery about your sleep habits?

YES NO

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You may keep the FitBit after you complete the study.

## **Additional Information**

NCT05044312 Protocol 2019-1182 May 14, 2020 

- 4. You may ask the study chair (Dr. Sriram Yennu, at 713-563-0034) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.

## **Future Research**

#### **Data**

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and/or shared with other researchers and/or institutions for use in future research.

## <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Study monitors and auditors who verify the accuracy of the information

Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

NCT05044312 Protocol 2019-1182 May 14, 2020 

#### CONSENT/AUTHORIZATION

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document. SIGNATURE OF PARTICIPANT DATE PRINTED NAME OF PARTICIPANT Medical Record Number **LEGALLY AUTHORIZED REPRESENTATIVE (LAR)** The following signature line should only be filled out when the participant does not have the capacity to legally consent to take part in the study and/or sign this document on his or her own behalf. SIGNATURE OF LAR DATE PRINTED NAME and RELATIONSHIP TO PARTICIPANT WITNESS TO CONSENT I was present during the explanation of the research to be performed under Protocol 2019-1182 SIGNATURE OF WITNESS TO THE VERBAL CONSENT DATE PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for vulnerable adult participants. If witnessing the assent of a pediatric participant, leave this line blank and sign on the witness to assent page instead.

PRINTED NAME OF WITNESS TO THE VERBAL CONSENT

## **PERSON OBTAINING CONSENT**

| representative, using language have fully informed this particip | study with the participant and/or his<br>e that is understandable and approp<br>pant of the nature of this study and i<br>ant understood this explanation. | riate. I believe that I |
|---|---|---|
| PERSON OBTAINING CONS | ENT | DATE |
| PRINTED NAME OF PERSON | N OBTAINING CONSENT | _ |
| subtractions) into(Na | me of Language)<br>ent by translating all questions and r | ed the people |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| ☐ Please check here if the translator was a member of the research team. (If checked, a witness, other than the translator, must sign the witness line below.) | | |
| SIGNATURE OF WITNESS TO COTHER THAN TRANSLATO OR STUDY CHAIR) | TO THE VERBAL TRANSLATION<br>OR, PARENT/GUARDIAN, | DATE |
| PRINTED NAME OF WITNES | S TO THE VERBAL TRANSLATION | |